CLINICAL TRIAL: NCT04583020
Title: Neoadjuvant PD-1 in Newly Diagnosed Glioblastoma: A Phase 2 Clinical Trial
Brief Title: Neoadjuvant PD-1 in Newly Diagnosed Glioblastoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS-2522
Record Dates: First submitted 2020-09-29; First posted 2020-10-12 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Glioblastoma
Keywords: Camrelizumab
MeSH Terms: conditions — Glioblastoma | interventions — camrelizumab; Radiation; Temozolomide

STUDY DESIGN:
Intervention Model Description: Neoadjuvant PD-1 inhibitor will be administered to patients with newly diagnosed glioblastomas, followed by surgical resection, standard radiochemotherapy, and further PD-1 inhibitor treatment
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Neoadjuvant PD-1 inhibitor (Experimental): Neoadjuvant PD-1 inhibitor Camrelizumab will be administered to patients with newly diagnosed glioblastomas, followed by surgical resection, standard radiochemotherapy, and further PD-1 inhibitor treatment.
  Interventions: Drug: Camrelizumab; Radiation: radiation; Drug: Temozolomide

INTERVENTIONS:
Drug: Camrelizumab — Neoadjuvant Camrelizumab 200mg IV, adjuvant Camrelizumab 200mg IV (once every two weeks, until progress)
Radiation: radiation — 60Gy/30
Drug: Temozolomide — Given PO during RT 75mg/m2/d; 4 weeks post RT 150-200mg/m2/d days 1-5, 4 weeks/cycle, 6 cycles
  Other Names: TMZ

SUMMARY:
The purpose of this research is to study the safety and efficacy of Camrelizumab treating patients with newly diagnosed glioblastomas.

DETAILED DESCRIPTION:
This is a phase II clinical trial. The purpose of this research is to study the safety and efficacy of Camrelizumab treating patients with newly diagnosed glioblastomas. Neoadjuvant PD-1 inhibitor will be administered to patients with newly diagnosed glioblastomas, followed by surgical resection, standard radiochemotherapy, and further PD-1 inhibitor treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be willing to provide informed consent.
2. Patient must be 18-70 years old.
3. Patient must be first diagnosed of WHO grade IV neural glioma by MRI, without previous treatment.
4. Patient must receive confine operation that can be delayed for at least 2 weeks, in order to receive neoadjuvant treatment; patient must not receive other antitumor therapy besides this study plan.
5. Karnofsky ≥ 70
6. If patient is on glucocorticoids treatment, the amount of glucocorticoids must be stable or decreasing at least 5 days before baseline MRI acquisition. Oral dexamethasone must be <3 tablets(0.75mg/tablet) at least 5 days before baseline MRI.
7. Patient has not received antibiotics for 1month before inclusion.
8. Estimate survival ≥12weeks.
9. Major organ functions normally, without severe blood, heart, lung, liver, renal abnormality or immune deficiency. Laboratory examination meets the following requirements:

   i. Complete blood count:
   1. HGB≥90g/L;
   2. WBC≥3.0×109/L, NEUT≥1.5×109/L;
   3. PLT ≥60×109/L;

   ii. Blood biochemistry:
   1. BIL≤1.5×upper limit of normal (ULN);
   2. ALT and AST≤2.0×ULN;
   3. Serum Cr≤1.5×ULN or Ccr≥50ml/min (Cockcroft-Gault formular);

   iii. Fecal occult blood(-);

   iv. Urine routines normal, or urine protein <(++), or 24h urine protein<1.0g;

   v. Left ventricular ejection fraction(LVEF)≥50%.
10. Normal clotting function, no active bleeding or thrombosis disease.

    1. INR≤1.5×ULN;
    2. APTT≤1.5×ULN;
    3. PT≤1.5ULN;
11. Female patients of childbearing potential must receive pregnancy test (serum or urine) with negative result, and voluntarily practice appropriate forms of contraception, during observation period and 8 weeks after final administration of Camrelizumab; male patients should receive surgical sterilization or agree to practice appropriate forms of contraception, during observation period and 8 weeks after final administration of Camrelizumab.
12. Patient should have good follow-up compliance.

Exclusion Criteria:

1. Patient with other malignant tumor history in five years (except complete treatment of cervical cancer in situ, basal cell carcinoma, squamous cell skin cancer).
2. Patient needs emergency surgery.
3. History of allergy to other monoclonal antibody or other ingredients; or can not receive MRI.
4. Previous immunotherapy (e.g. PD-1, PD-L1, CTLA-4), previous intracranial radiotherapy.
5. Any previous investigational medication within 4 weeks before first administration of Camrelizumab.
6. Included in another clinical investigation simultaneously, except for observational (non-interventional) clinical study or follow-up of an interventional clinical study.
7. Already has meningioma, multiple gliomas, extracranial lesions. The definition of multiple gliomas is: discontinuous strong signal on T2/FLAIR; satellite lesions.
8. History of antitumor vaccine injection, or history of live vaccine injection within 4 weeks before first administration of Camrelizumab.
9. Less than 4 weeks after the latest surgery, radiochemotherapy, glucocorticoids treatment, immunotherapy, targeted therapy.
10. Thrombosis event within 12 months before inclusion, such as cerebrovascular accident (TIA, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, pulmonary embolism.
11. Any unstable systematic disease (including active infection, uncontrolled hypertension, unstable angina, medical treatment needed liver, kidney, metabolic disease).
12. Heart failure with NYHA grade 2 or above, unstable angina, myocardial infarction within 1 year, treatment needed supraventricular or ventricular arrhythmia.
13. Patient with known HIV infection or active hepatitis.
14. History or risk of autoimmune disease, such as systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, glomerulonephritis. Patient is allowed to be included, if eczema, psoriasis or leukoderma is well controlled at baseline, with only local weak steroid treatment.
15. Systematic immune suppressor, such as prednisone, cyclophosphamide, amethopterin, azathioprim, thalidomide, anti-TNF drugs. Low dose of systematic immune suppressor is allowed (e.g. single dose of dexamethasone for nausea). Patient with postural hypotension or adrenocortical insufficiency is allowed to use inhaled corticosteroids and mineralocorticoid.
16. History of interstitial lung disease, idiopathic pulmonary fibrosis, pneumonia, tissue pneumonia, or evidence of active pneumonia on CT scan. Radiation pneumonia or pulmonary fibrosis is allowed in patient with radiation history.
17. Other chronic disease that requires immune suppressor or corticosteroids treatment.
18. Female patients who are pregnant or currently breastfeeding.
19. Active infection or fever of unknown origin >38.5℃ at the first administration of Camrelizumab.
20. Blood clotting abnormality, bleeding tendency or receiving thrombolytic or anticoagulant therapy.
21. Patient with known history of Psychotropic drug abuse, alcoholism or drug addiction.
22. Other situation determined by the researcher that may influence the conduction or result of the clinical study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2020-11-12 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | up to 12 months
  Survival will be assessed at 6 months and 12 months from the time of recruitment until the time of death. Kaplan-Meier survival analyses will be performed.
Progression-free survival (PFS) | up to 12 months
  Progression-free survival will be assessed at 6 months and 12 months from the time of recruitment until the time of death. Kaplan-Meier survival analyses will be performed.

SECONDARY OUTCOMES:
Proportion of participants with treatment-related adverse events | up to 2 years
  toxicity assessed by Common Toxicity Criteria (CTC) version
Objective response rate (ORR) | up to 2 years
  response rate assessed by Response Assessment in Neuro-Oncology (RANO) criteria

CONTACTS AND LOCATIONS:
Overall Officials: Yu Wang, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
There is no IPD share plan.